CLINICAL TRIAL: NCT01347580
Title: A 30 Day International, Randomized, Parallel-group, Double-blind, Placebo-controlled Phase IV Study to Evaluate Efficacy and Safety of Pre-hospital vs. In-hospital Initiation of Ticagrelor Therapy in STEMI Patients Planned for PCI.
Brief Title: A 30 Day Study to Evaluate Efficacy and Safety of Pre-hospital vs. In-hospital Initiation of Ticagrelor Therapy in STEMI Patients Planned for Percutaneous Coronary Intervention (PCI)
Acronym: ATLANTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5130L00006
Record Dates: First submitted 2011-04-19; First posted 2011-05-04 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Myocardial Infarction; Segment Elevation Myocardial Infarction (STEMI)
Keywords: Heart attack; heart disease; cardiovascular disease; stroke; reperfusion; pre hospital settings; ticagrelor; Percutaneous Coronary Intervention
MeSH Terms: conditions — Myocardial Infarction; Heart Diseases; Cardiovascular Diseases; Stroke | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Loading dose of Ticagrelor (180 mg) followed by matching placebo. After the loading dose the patient will receive Ticagrelor (90 mg bid) for 30 days.
  Interventions: Drug: Ticagrelor
- Placebo (Experimental): Placebo followed by a loading dose of Ticagrelor (180 mg). After the loading dose the patient will receive Ticagrelor (90 mg bid) for 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ticagrelor — Oral Ticagrelor loading dose (180 mg) followed by matching placebo
  Arms: Ticagrelor
Drug: Placebo — Placebo followed by oral Ticagrelor loading dose (180 mg)
  Arms: Placebo

SUMMARY:
The aim of this study is to determine whether initiation of ticagrelor as early as in the ambulance setting leads to a rapid reperfusion of the infarct-related artery therefore facilitating the Percutaneous Coronary Intervention (PCI) and optimizing the outcome for the patient.

The study will assess the efficacy and safety of pre-hospital compared to in-hospital administration of ticagrelor in co-administration with aspirin, on restoring the blood flow in the occluded heart artery and improving the myocardial perfusion in patients suffering from myocardial infarction and planned to have a PCI. Patients can be randomised in either one of the 2 arms:

re-hospital ticagrelor arm: Patients will receive a loading dose of 180 mg ticagrelor for the pre-hospital administration and placebo for in-hospital administration.

or In-hospital ticagrelor arm: Patients will receive a placebo for pre-hospital administration and 180 mg ticagrelor loading dose for in-hospital administration.

Patients are initially managed by ambulance physician/personnel in pre hospital settings. They are then transferred into a Catheterization room to undergo a PCI.

After the administration of the loading dose of ticagrelor (double blind), patients will continue on ticagrelor 90 mg bid and be followed in study for 30 days post randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Women must not be of child-bearing potential (1 year post-menopausal or surgically sterile).
* Symptoms of acute MI of more than 30 min but less than 6 hours
* New persistent ST-segment elevation ≥ 1 mm in two or more contiguous electrocardiogram (ECG) leads.

Exclusion Criteria:

* Expected time to 1st PCI balloon inflation in the hospital, from the qualifying ECG is more than 120 minutes
* Contraindication to ticagrelor (refer to SmPC)
* Concomitant medication that may increase the risk of bleeding [e.g non steroidal anti-inflammatory drugs (NSAIDs), oral anticoagulant and / or fibrinolytics, planned or administered 24 hours before randomization]
* Any of the following conditions in the absence of a functioning implanted pacemaker: known SSS, second or third degree AVB, or documented syncope of suspected bradycardic origin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1875 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Judith Hsia, MD, Study Director — AstraZeneca; Pr Gilles Montalescot, Principal Investigator — Pitie Salpetriere Hospital
Locations (96):
- Algeria (2):
  - Research Site, Algiers
  - Research Site, Blida
- Australia (3):
  - Research Site, Herston
  - Research Site, Southport
  - Research Site, Woolloongabba
- Austria (3):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Vienna
- Canada (4):
  - Research Site, Halifax, Nova Scotia
  - Research Site, Newmarket, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Regina, Saskatchewan
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Odense C
- France (28):
  - Research Site, Aubervilliers
  - Research Site, Besançon
  - Research Site, Boulogne-Billancourt
  - Research Site, Bourges
  - Research Site, Bron
  - Research Site, Châteauroux
  - Research Site, Corbeil-Essonnes
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Lagny-sur-Marne
  - Research Site, Le Chesnay
  - Research Site, Le Coudray
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Massy
  - Research Site, Melun
  - Research Site, Montauban
  - Research Site, Montfermeil
  - Research Site, Montreuil
  - Research Site, Neuilly-sur-Seine
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Quincy-sous-Sénart
  - Research Site, Rouen
  - Research Site, Strasbourg
  - Research Site, Tours
  - Research Site, Vannes
- Germany (12):
  - Research Site, Bad Friedrichshall
  - Research Site, Bad Nauheim
  - Research Site, Darmstadt
  - Research Site, Esslingen am Neckar
  - Research Site, Freiburg im Breisgau
  - Research Site, Giessen
  - Research Site, Hanover
  - Research Site, Ludwigshafen
  - Research Site, Lüdenscheid
  - Research Site, Mainz
  - Research Site, Merseburg
  - Research Site, Wuppertal
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Pécs
  - Research Site, Szeged
- Italy (9):
  - Research Site, Arezzo
  - Research Site, Ascoli Piceno
  - Research Site, Cona
  - Research Site, Forlì
  - Research Site, Genova
  - Research Site, Grosseto
  - Research Site, Massa
  - Research Site, Seriate
  - Research Site, Siena
- Netherlands (4):
  - Research Site, 's-Hertogenbosch
  - Research Site, Alkmaar
  - Research Site, Arnhem
  - Research Site, Terneuzen
- Spain (10):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Hospitalet de Llobregat(Barcel
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville
  - Research Site, Vigo(Pontevedra)
- Sweden (4):
  - Research Site, Gävle
  - Research Site, Linköping
  - Research Site, Örebro
  - Research Site, Uppsala
- United Kingdom (10):
  - Research Site, Ashford
  - Research Site, Belfast
  - Research Site, Cambridge
  - Research Site, Coventry
  - Research Site, Eastbourne
  - Research Site, Hastings
  - Research Site, Middlesbrough
  - Research Site, Newcastle upon Tyne
  - Research Site, Norwich
  - Research Site, Sheffield

REFERENCES:
- [Result] Montalescot G, van 't Hof AW, Lapostolle F, Silvain J, Lassen JF, Bolognese L, Cantor WJ, Cequier A, Chettibi M, Goodman SG, Hammett CJ, Huber K, Janzon M, Merkely B, Storey RF, Zeymer U, Stibbe O, Ecollan P, Heutz WM, Swahn E, Collet JP, Willems FF, Baradat C, Licour M, Tsatsaris A, Vicaut E, Hamm CW; ATLANTIC Investigators. Prehospital ticagrelor in ST-segment elevation myocardial infarction. N Engl J Med. 2014 Sep 11;371(11):1016-27. doi: 10.1056/NEJMoa1407024. Epub 2014 Sep 1. PMID 25175921
- [Derived] Lapostolle F, Van't Hof AW, Hamm CW, Stibbe O, Ecollan P, Collet JP, Silvain J, Lassen JF, Heutz WMJM, Bolognese L, Cantor WJ, Cequier A, Chettibi M, Goodman SG, Hammett CJ, Huber K, Janzon M, Merkely B, Storey RF, Ten Berg J, Zeymer U, Licour M, Tsatsaris A, Montalescot G; ATLANTIC Investigators. Morphine and Ticagrelor Interaction in Primary Percutaneous Coronary Intervention in ST-Segment Elevation Myocardial Infarction: ATLANTIC-Morphine. Am J Cardiovasc Drugs. 2019 Apr;19(2):173-183. doi: 10.1007/s40256-018-0305-0. PMID 30353444
- [Derived] Fabris E, Van't Hof A, Hamm CW, Lapostolle F, Lassen JF, Goodman SG, Ten Berg JM, Bolognese L, Cequier A, Chettibi M, Hammett CJ, Huber K, Janzon M, Merkely B, Storey RF, Zeymer U, Cantor WJ, Kerneis M, Diallo A, Vicaut E, Montalescot G; ATLANTIC investigators. Pre-hospital administration of ticagrelor in diabetic patients with ST-elevation myocardial infarction undergoing primary angioplasty: A sub-analysis of the ATLANTIC trial. Catheter Cardiovasc Interv. 2019 Jun 1;93(7):E369-E377. doi: 10.1002/ccd.27921. Epub 2018 Oct 9. PMID 30302940
- [Derived] Bagai A, Goodman SG, Cantor WJ, Vicaut E, Bolognese L, Cequier A, Chettibi M, Hammett CJ, Huber K, Janzon M, Lapostolle F, Lassen JF, Merkely B, Storey RF, Ten Berg JM, Zeymer U, Diallo A, Hamm CW, Tsatsaris A, El Khoury J, Van't Hof AW, Montalescot G. Duration of ischemia and treatment effects of pre- versus in-hospital ticagrelor in patients with ST-segment elevation myocardial infarction: Insights from the ATLANTIC study. Am Heart J. 2018 Feb;196:56-64. doi: 10.1016/j.ahj.2017.10.021. Epub 2017 Nov 4. PMID 29421015
- [Derived] Kilic S, Fabris E, Van't Hof AWJ, Hamm CW, Lapostolle F, Lassen JF, Tsatsaris A, Diallo A, Vicaut E, Montalescot G; ATLANTIC Investigators. Thrombus aspiration and prehospital ticagrelor administration in ST-elevation myocardial infarction: Findings from the ATLANTIC trial. Am Heart J. 2018 Feb;196:1-8. doi: 10.1016/j.ahj.2017.09.018. Epub 2017 Oct 3. PMID 29421001
- [Derived] Venetsanos D, Sederholm Lawesson S, Alfredsson J, Janzon M, Cequier A, Chettibi M, Goodman SG, Van't Hof AW, Montalescot G, Swahn E. Association between gender and short-term outcome in patients with ST elevation myocardial infraction participating in the international, prospective, randomised Administration of Ticagrelor in the catheterisation Laboratory or in the Ambulance for New ST elevation myocardial Infarction to open the Coronary artery (ATLANTIC) trial: a prespecified analysis. BMJ Open. 2017 Sep 21;7(9):e015241. doi: 10.1136/bmjopen-2016-015241. PMID 28939567
- [Derived] Cayla G, Lapostolle F, Ecollan P, Stibbe O, Benezet JF, Henry P, Hammett CJ, Lassen JF, Storey RF, Ten Berg JM, Hamm CW, Van't Hof AW, Montalescot G; ACTION study group. Pre-hospital ticagrelor in ST-segment elevation myocardial infarction in the French ATLANTIC population. Int J Cardiol. 2017 Oct 1;244:49-53. doi: 10.1016/j.ijcard.2017.06.009. Epub 2017 Jun 9. PMID 28622941
- [Derived] Lupi A, Schaffer A, Lazzero M, Tessitori M, De Martino L, Rognoni A, Bongo AS, Porto I. Pre-hospital ticagrelor in patients with ST-segment elevation myocardial infarction with long transport time to primary PCI facility. Cardiovasc Revasc Med. 2016 Dec;17(8):528-534. doi: 10.1016/j.carrev.2016.08.005. Epub 2016 Aug 20. PMID 27666002
- [Derived] Silvain J, Storey RF, Cayla G, Esteve JB, Dillinger JG, Rousseau H, Tsatsaris A, Baradat C, Salhi N, Hamm CW, Lapostolle F, Lassen JF, Collet JP, Ten Berg JM, Van't Hof AW, Montalescot G. P2Y12 receptor inhibition and effect of morphine in patients undergoing primary PCI for ST-segment elevation myocardial infarction. The PRIVATE-ATLANTIC study. Thromb Haemost. 2016 Aug 1;116(2):369-78. doi: 10.1160/TH15-12-0944. Epub 2015 May 19. PMID 27196998
- [Derived] Montalescot G, van 't Hof AW, Bolognese L, Cantor WJ, Cequier A, Chettibi M, Collet JP, Goodman SG, Hammett CJ, Huber K, Janzon M, Lapostolle F, Lassen JF, Licour M, Merkely B, Salhi N, Silvain J, Storey RF, Ten Berg JM, Tsatsaris A, Zeymer U, Vicaut E, Hamm CW; ATLANTIC Investigators. Effect of Pre-Hospital Ticagrelor During the First 24 h After Primary Percutaneous Coronary Intervention in Patients With ST-Segment Elevation Myocardial Infarction: The ATLANTIC-H(2)(4) Analysis. JACC Cardiovasc Interv. 2016 Apr 11;9(7):646-56. doi: 10.1016/j.jcin.2015.12.024. Epub 2016 Mar 5. PMID 26952907
- [Derived] Montalescot G, Lassen JF, Hamm CW, Lapostolle F, Silvain J, ten Berg JM, Cantor WJ, Goodman SG, Licour M, Tsatsaris A, van't Hof AW. Ambulance or in-catheterization laboratory administration of ticagrelor for primary percutaneous coronary intervention for ST-segment elevation myocardial infarction: rationale and design of the randomized, double-blind Administration of Ticagrelor in the cath Lab or in the Ambulance for New ST elevation myocardial Infarction to open the Coronary artery (ATLANTIC) study. Am Heart J. 2013 Apr;165(4):515-22. doi: 10.1016/j.ahj.2012.12.015. Epub 2013 Feb 13. PMID 23537967
- See also: D5130L00006_Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=482&filename=D5130L00006_Protocol_Redacted.pdf
- See also: D5130L00006_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=482&filename=D5130L00006_CSR_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized in pre-hospital settings at 102 Emergency Medical Services between September 2011 and October 2013. 1875 patients were recruited in the study, 1862 consented patients were randomized.
Groups:
- Pre-hospital Ticagrelor: Loading dose of Ticagrelor (180 mg) followed by matching placebo. After the loading dose the patient will receive Ticagrelor (90 mg bid) for 30 days.
- In-hospital Ticagrelor: Placebo followed by a loading dose of Ticagrelor (180 mg). After the loading dose the patient will receive Ticagrelor (90 mg bid) for 30 days.
Period: Overall Study
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Started | 909 (based on randomized treatment) | 953 (based on randomized treatment)
Modified Intent to Treat Population | 906 (based on randomized treatment) | 952 (based on randomized treatment)
Safety Population | 908 (based on actual treatment) | 950 (based on actual treatment)
Completed | 844 (based on randomized treatment) | 897 (based on randomized treatment)
Not Completed | 65 | 56
Not completed — Withdrawal by Subject | 13 | 23
Not completed — Death | 30 | 19
Not completed — Protocol Violation | 10 | 7
Not completed — Lost to Follow-up | 3 | 1
Not completed — Had other reason | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor | Total
Number analyzed (Participants) | 909 | 953 | 1862
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 60.6 (12.38) | 61.0 (12.49) | 60.8 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 196 | 369
  Male | 736 | 757 | 1493
Diabetes mellitus [Number; unit: patients]
  yes | 115 | 138 | 253
  no/unknown | 794 | 815 | 1609
TIMI risk score [Number; unit: patients] — Thrombolysis in Myocardial Infarction (TIMI) is a scoring system based on independant predictors of mortality such as age, diabetes mellitus, history of hypertension, history of angina, ST segment elevation. The death rate at 30 days for the following scores are: 0-2: 0.8%-2.2%, 3-6: 4.4% -16.1%, score>6: 23.4% to 35.9%.
  patients
    0-2 | 552 | 573 | 1125
    3-6 | 337 | 365 | 702
    >6 | 20 | 15 | 35
Killip class [Number; unit: patients] — Killip class assesses the presence and severity of heart failure by physical examination. Class I :No rales, no 3rd heart sound. Class 2: Rales in <1⁄2 lung field or presence of a 3rd heart sound. Class 3: Rales in >1⁄2 lung field-pulmonary edema.Class 4 : Cardiogenic shock-determined clinically.
  patients
    I | 819 | 862 | 1681
    II, III, IV | 51 | 43 | 94
    unknown | 39 | 48 | 87
First medical contact [Number; unit: patients]
  in ambulance | 689 | 723 | 1412
  in emergency department | 220 | 230 | 450
PCI [Number; unit: Patients] — Percutaneous coronary intervention (PCI) is a non-surgery intervention performed to open blocked coronary arteries and to restore arterial blood flow to the heart tissue.
  Patients
    yes | 800 | 830 | 1630
    no | 109 | 123 | 232
type of PCI [Number; unit: patients] — on patients with PCI
  patients
    with stent | 760 | 776 | 1536
    without stent | 40 | 54 | 94
Time between the 2 loading doses [Median (Inter-Quartile Range); unit: minutes] | 32 [22 to 45] | 30 [22 to 43] | 31 [22 to 44]

OUTCOME MEASURES:

1. Primary Outcome: Thrombolysis In Myocardial Infarction (TIMI) Flow Grade 3 of MI Culprit Vessel at Initial Angiography (Co-primary Endpoint)
Description: (TIMI) flow grade classification is used to assess coronary blood flow in acute coronary syndromes. grade 0:no reperfusion, grade 1: penetration without perfusion, grade 2: Partial reperfusion, grade 3: complete perfusion.
Time Frame: At initial angiography, pre PCI
Population: mITT, on patients with non missing values
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 824 | 856
patients | 143 | 145
Statistical Analysis 1: Comparison: Pre-hospital Ticagrelor vs In-hospital Ticagrelor; Test type: Superiority or Other; p = 0.8214, Regression, Logistic — pvalue at 0.025 , adjusted for multiple comparisons; Odds Ratio (OR) = 1.030, 95% CI 2-sided [0.799 to 1.327]

2. Primary Outcome: ST-segment Elevation Resolution Pre PCI ≥70% (Co-primary Endpoint)
Description: ST segment elevation resolution is the mean ST elevation pre-hospital minus the mean STelevation pre-PCI divided by the mean ST elevation pre-hospital. It is expressed as a percentage and split in 2 categories , complete (≥70%) versus incomplete (<70%) resolution.
Time Frame: Between baseline and PCI
Population: mITT, on patients with non missing values
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 774 | 824
patients | 102 | 102
Statistical Analysis 1: Comparison: Pre-hospital Ticagrelor vs In-hospital Ticagrelor; Test type: Superiority or Other; p = 0.6322, Regression, Logistic — P value at 0.025 adjusted for multiple comparisons; Odds Ratio (OR) = 1.074, 95% CI 2-sided [0.801 to 1.441]

3. Secondary Outcome: 1st Composite Clinical Endpoint
Description: death/MI/stroke/urgent revascularization/stent thrombosis. Adjudicated events except death
Time Frame: during the 30 days of treatment
Population: mITT
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 906 | 952
patients | 41 | 42
Statistical Analysis 1: Comparison: Pre-hospital Ticagrelor vs In-hospital Ticagrelor; Test type: Superiority or Other; p = 0.9056, Regression, Logistic; Odds Ratio (OR) = 1.027, 95% CI 2-sided [0.661 to 1.595]

4. Secondary Outcome: 2nd Composite Clinical Endpoint
Description: Death/MI/urgent revascularization. Adjudicated events except death
Time Frame: within 30 days of study
Population: mITT
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 906 | 952
patients | 39 | 34
Statistical Analysis 1: Comparison: Pre-hospital Ticagrelor vs In-hospital Ticagrelor; Test type: Superiority or Other; p = 0.4168, Regression, Logistic; Odds Ratio (OR) = 1.215, 95% CI 2-sided [0.760 to 1.942]

5. Secondary Outcome: Definite Stent Thrombosis
Description: Definite stent thrombosis is considered to have occurred by either angiographic or pathologic confirmation. It is an adjudicated endpoint
Time Frame: during 30 days of treatment
Population: mITT
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 906 | 952
patients | 2 | 11
Statistical Analysis 1: Comparison: Pre-hospital Ticagrelor vs In-hospital Ticagrelor; Test type: Superiority or Other; p = 0.0307, Regression, Logistic; Odds Ratio (OR) = 0.189, 95% CI 2-sided [0.042 to 0.856]

6. Secondary Outcome: TIMI Flow Grade 3 Post -PCI
Description: TIMI) flow grade 3 is complete perfusion post-PCI.
Time Frame: at coroangiography post-PCI
Population: mITT, on patients with non missing TIMI flow grade values
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 760 | 784
patients | 625 | 630
Statistical Analysis 1: Comparison: Pre-hospital Ticagrelor vs In-hospital Ticagrelor; Test type: Superiority or Other; p = 0.344, Regression, Logistic; Odds Ratio (OR) = 1.132, 95% CI 2-sided [0.876 to 1.462]

7. Secondary Outcome: ST Segment Elevation Resolution Post-PCI >= 70%
Description: ST segment elevation resolution post PCI >=70% is defined as complete resolution
Time Frame: Between baseline and ECG 60 mn post-PCI
Population: mITT on patients with non missing ECG values
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 713 | 743
patients | 410 | 390
Statistical Analysis 1: Comparison: Pre-hospital Ticagrelor; Test type: Superiority or Other; p = 0.0547, Regression, Logistic; Odds Ratio (OR) = 1.225, 95% CI 2-sided [0.996 to 1.506]

8. Secondary Outcome: Thrombotic Bail-out With GPIIb/IIIa Inhibitors at Initial PCI
Description: Glycoprotein (GP) IIb/IIIa inhibitors are often used as a rescue or bailout therapy to manage complications arising during percutaneous coronary intervention.
Time Frame: during PCI
Population: mITT
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 906 | 952
patients | 78 | 100
Statistical Analysis 1: Comparison: Pre-hospital Ticagrelor vs In-hospital Ticagrelor; Test type: Superiority or Other; p = 0.1660, Regression, Logistic; Odds Ratio (OR) = 0.803, 95% CI 2-sided [0.588 to 1.096]

9. Secondary Outcome: Major Bleeds Within 48 Hours
Description: non CABG related bleeds, (PLATO definition) include Life threatening and other major bleeds
Time Frame: within 48 hours of first dose
Population: Safety
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 908 | 950
patients | 16 | 15

10. Secondary Outcome: Minor and Major Bleedings Within 48 Hours
Description: non CABG related bleeds (PLATO definition)
Time Frame: within 48 hours of first dose
Population: Safety
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 908 | 950
patients | 24 | 24

11. Secondary Outcome: Major Bleeds After 48 Hours
Description: non CABG related bleeds (PLATO definition) include life threatening and other major bleedings
Time Frame: after 48hours post-first dose
Population: safety
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 908 | 950
patients | 11 | 11

12. Secondary Outcome: Minor and Major Bleeds After 48 Hours
Description: non CABG related bleeds (PLATO definition)
Time Frame: after 48 hours post first dose
Population: safety
Measure: Number; unit: patients
Arm/Group | Pre-hospital Ticagrelor | In-hospital Ticagrelor
Number analyzed (Participants) | 908 | 950
patients | 18 | 16

ADVERSE EVENTS:
Time Frame: within 30 days of study
Description: Actual Treatment Safety analysis set concerns 1858 patients - Ticagrelor pre-hosp:908 and Ticagrelor in-hosp: 950. 4 patients receiveived study medication not according to randomization assignment
Groups:
- Ticagrelor In-Hosp: Placebo followed by a loading dose of Ticagrelor (180 mg). After the loading dose the patient will receive Ticagrelor (90 mg bid) for 30 days.
- Ticagrelor Pre-Hosp: Loading dose of Ticagrelor (180 mg) followed by matching placebo. After the loading dose the patient will receive Ticagrelor (90 mg bid) for 30 days.
Arm/Group | Ticagrelor In-Hosp | Ticagrelor Pre-Hosp
Serious Adverse Events (participants affected / at risk) | 143/950 | 140/908
Other Adverse Events (participants affected / at risk) | 529/950 | 469/908
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor In-Hosp (N=950) | Ticagrelor Pre-Hosp (N=908)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 2 (2) | 3 (3)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 1 (1)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 1 (1)
ARTERIOSPASM CORONARY (Cardiac disorders) | 2 (2) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 4 (4)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 3 (3) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 2 (2) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 7 (7) | 11 (11)
CARDIAC ASTHMA (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 7 (7) | 7 (7)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 2 (2)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOGENIC SHOCK (Cardiac disorders) | 16 (16) | 17 (17)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 1 (1)
DRESSLER'S SYNDROME (Cardiac disorders) | 1 (1) | 2 (2)
INTERVENTRICULAR SEPTUM RUPTURE (Cardiac disorders) | 1 (1) | 0 (0)
INTRACARDIAC THROMBUS (Cardiac disorders) | 4 (4) | 2 (2)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 2 (2)
MYOCARDIAL RUPTURE (Cardiac disorders) | 1 (1) | 1 (1)
PALPITATIONS (Cardiac disorders) | 2 (2) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 4 (4) | 0 (0)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
TORSADE DE POINTES (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICLE RUPTURE (Cardiac disorders) | 1 (1) | 1 (1)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 30 (30) | 23 (23)
VENTRICULAR SEPTAL DEFECT ACQUIRED (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 7 (7) | 6 (6)
VENTRICULAR SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTROINTESTINAL TELANGIECTASIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 1 (1) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 2 (2)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
CARDIAC DEATH (General disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 4 (4) | 1 (1)
DEVICE MALFUNCTION (General disorders) | 0 (0) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 2 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 5 (5) | 4 (4)
SUDDEN CARDIAC DEATH (General disorders) | 1 (1) | 0 (0)
SUDDEN DEATH (General disorders) | 1 (1) | 2 (2)
THROMBOSIS IN DEVICE (General disorders) | 1 (1) | 0 (0)
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 0 (0) | 1 (1)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 2 (2)
BILIARY SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
GROIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 2 (2)
RELAPSING FEVER (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1)
NUTRITIONAL CONDITION ABNORMAL (Investigations) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
TROPONIN INCREASED (Investigations) | 0 (0) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ADRENAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CARDIAC MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
EXTRANODAL MARGINAL ZONE B-CELL LYMPHOMA (MALT TYPE) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RECTAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RENAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 (2) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 1 (1)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 3 (3) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 2 (2)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 2 (2)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DIAPHRAGMATIC PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
AORTIC DISSECTION (Vascular disorders) | 1 (1) | 2 (2)
ARTERY DISSECTION (Vascular disorders) | 2 (2) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor In-Hosp (N=950) | Ticagrelor Pre-Hosp (N=908)
Ventricular tachycardia (Cardiac disorders) | 81 | 79
Dyspnoea (Gastrointestinal disorders) | 86 | 62
Nausea (Gastrointestinal disorders) | 49 | 41
Non cardiac chest pain (General disorders) | 52 | 42
Hypotension (Vascular disorders) | 30 | 44
Hypokalaemia (Metabolism and nutrition disorders) | 26 | 28
Headache (Nervous system disorders) | 31 | 19
Vomiting (Gastrointestinal disorders) | 40 | 34
Atrial fibrillation (Cardiac disorders) | 38 | 30
Ventricular fibrillation (Cardiac disorders) | 37 | 32
Cardiac failure (Cardiac disorders) | 33 | 30
Bradycardia (Cardiac disorders) | 26 | 28

LIMITATIONS AND CAVEATS:
This urgent setting study included 8.6% of patients with symptoms of MI in ambulance but having finally not a STEMI diagnosis in cathlab.

No prespecified hypothesis and procedure for adjustment was made on secondary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less